CLINICAL TRIAL: NCT01429883
Title: Extracorporeal Shock Wave Treatment - Can the Pain be Reduced?
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ESWTRUZ01
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Fasciitis, Plantar; Achillodynia; Periarthritis Calcarea; Epikondylopathia Humeri /Radii
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with Fascititis plantaris, Achillodynie, Periarthropathia humerosacpularis calcarea or Epikondylopathia humeri /radii get the shock wave therapy in our clinic as planned. During our study the investigators want to ask for pain, pain reduction and function.

DETAILED DESCRIPTION:
Patients with either Fascititis plantaris, Achillodynie, Periarthropathia humerosacpularis calcarea or Epikondylopathia humeri /radii get a shock wave therapy in our clinic of rheumatology as planned. During our study the investigators ask for pain, pain reduction and function (all questionnaires).

ELIGIBILITY:
Inclusion criteria:

-Patients with:

* Fascititis plantaris,
* Achillodynie,
* Periarthropathia humerosacpularis calcarea or
* Epicondylopathia humeri /radii, who got the shock wave therapy.

Exclusion criteria:

* Anticoagulation,
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Fascititis plantaris, Achillodynie, Periarthropathia humerosacpularis calcarea or Epikondylopathia humeri /radii, who got the shock wave therapy.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Sandra Blumhardt, MD, Principal Investigator — University Hospital Zurich, Division of Rheumatology
Locations (1):
- University Hospital, Zurich, Switzerland